CLINICAL TRIAL: NCT04565808
Title: CHA2DS2-VASc Score as a Predictor of Thrombus Burden, No-Reflow Phenomenon and Clinical Outcomes in Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: CHA2DS2-VASc Score as a Predictor of Thrombus Burden and Clinical Outcomes in Patients Undergoing PPCI.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osman Ahmed Osman Ahmed, Doctor, Assiut University
Other Study IDs: CHA2DS2-VASc Score in PPCI
Record Dates: First submitted 2020-09-16; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: primary percutaneous coronary intervention — Primary Percutaneous Coronary Intervention (PPCI), also known as angioplasty or coronary angioplasty, is a procedure used to diagnose and treat the narrowed coronary arteries of the heart.
  Other Names: coronary angioplasty

SUMMARY:
Aim of the work is to evaluate the use CHA2DS2-VASc score in predicting no-reflow phenomenon and its impact on short term primary percutaneous coronary intervention outcomes (in-hospital mortality) and long term (6 months) incidence of MACE ( major adverse cardiac event ) in patients with ST segment elevation Myocardial infarction who underwent primary primary percutaneous coronary intervention

DETAILED DESCRIPTION:
Large intracoronary thrombus burden is known to be associated with reduced procedural success during the Primary Percutaneous Coronary Intervention (PPCI), larger infarct size, increased ischemic complications and mortality. No-Reflow phenomenon is related to higher incidence of complications, and short- and long-term morbidity and mortality in acute STEMI patients.

Although many risk factors were suggested, Tragically there's no widely accepted risk stratification method to anticipate these complications.

CHA2DS2-VASc score is a sum of several risk factors for thromboembolism. It is considered a clinical indicator of thromboembolic diseases and is recommended by the current guidelines for the estimation of thromboembolic events in patients with atrial fibrillation.

In this study, we evaluate the use CHA2DS2-VASc score as a novel rapid simple tool for predicting No-reflow and clinical outcomes among patients with STEMI who underwent primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with STEMI and undergoing primary Primary percutaneous coronary intervention.
* Patient Loaded pre-procedural with using with Aspirin 300 mg plus Ticagrelor 180 mg or Clopidogrel 600 mg.

Exclusion Criteria:

* Patients with chest pain more than 48 hours
* Patients not eligible for primary PCI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who are diagnosed as STEMI and undergoing primary PCI in Assiut University hospitals, Cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
TIMI (Thrombolysis in myocardial infarction) flow after Primary Percutaneous Coronary Intervention (No-reflow phenomenon versus normal flow) | Baseline
  Evaluation of the use of CHA2DS2-VASc score in predicting no-reflow phenomenon in patients with ST segment elevation myocardial infarction and undergoing Primary Percutaneous Coronary Intervention

SECONDARY OUTCOMES:
Early in-hospital complications and in-hospital mortality. | In-hospital stay duration ( up to 72 hours after intervention)
  Evaluation of the use of CHA2DS2-VASc score in predicting In-hospital incidence of MACE (including cardiovascular death, myocardial infarction, hospitalization because of heart failure and ischemic stroke)
Six months follow up | Six months follow up after hospital discharge
  Evaluation of the use of CHA2DS2-VASc score in predicting incidence of major adverse cardiovascular events which includes cardiovascular death, myocardial infarction, hospitalization because of heart failure and ischemic stroke during a Follow up period of 180 days after undergoing PPCI.

REFERENCES:
- [Background] Durante A, Camici PG. Novel insights into an "old" phenomenon: the no reflow. Int J Cardiol. 2015;187:273-80. doi: 10.1016/j.ijcard.2015.03.359. Epub 2015 Mar 26. PMID 25838230
- [Background] Goto K, Lansky AJ, Nikolsky E, Fahy M, Feit F, Ohman EM, White HD, Mehran R, Bertrand ME, Desmet W, Hamon M, Stone GW. Prognostic significance of coronary thrombus in patients undergoing percutaneous coronary intervention for acute coronary syndromes: a subanalysis of the ACUITY (Acute Catheterization and Urgent Intervention Triage strategY) trial. JACC Cardiovasc Interv. 2011 Jul;4(7):769-77. doi: 10.1016/j.jcin.2011.02.019. PMID 21777885